CLINICAL TRIAL: NCT00002252
Title: A Multicenter Placebo-Controlled Dose Titration Study to Evaluate the Efficacy and Safety of Sandostatin (SMS 201-995) in the Treatment of Patients With Acquired Immunodeficiency Related Diarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sandoz (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 102A; D203
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-08

CONDITIONS: Diarrhea; HIV Infections
Keywords: Octreotide; Diarrhea; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — Diarrhea; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Octreotide

INTERVENTIONS:
Drug: Octreotide

SUMMARY:
To determine the efficacy and safety of Sandostatin (octreotide) compared to placebo in controlling diarrhea which is a manifestation or complication of documented HIV infection and which is refractory (does not respond) to all known treatment classes.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Uncontrolled diarrhea that is either a manifestation or complication of documented HIV infection.
* Ability to communicate, participate, and comply with the requirements of the study.
* Capability of self administering injections of study medication or have responsible family member or companion who can.
* Given written consent prior to study entry.

Prior Medication:

Required:

* At least two weeks of conventional dosing regimens of antidiarrheal medication (e.g.:
* Lomotil, Imodium, Paregoric) within one month prior to study entry. OR Patients with evidence of upper or lower GI infection(s) for which there is approved, potentially curative therapy must have failed appropriate treatment for at least two weeks.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Evidence of underlying immunosuppressive disease other than due to HIV.
* Diarrhea caused by a known gastrointestinal disorder such as idiopathic ulcerative colitis, Crohn's disease, acute stool culture positive bacterial colitis (documented within the last 2 weeks prior to study entry AND not having at least 2 weeks of antibiotic therapy), pseudomembranous colitis (Clostridium difficile toxin positive), short gut syndrome, chronic pancreatitis (alcoholic or idiopathic), ischemic bowel disease, or enteroenteric fistulae.

Patients with the following are excluded:

* Diarrhea that can be controlled with conventional antidiarrheal agents.
* Stool weight at either of the 2 baseline periods that average < 500 g/day.
* Evidence of underlying immunosuppressive disease other than due to HIV.
* Diarrhea caused by other gastrointestinal disorders not related to HIV.

Prior Medication:

Excluded:

* Previously treated with Sandostatin as an anti-diarrheal agent.
* Experimental antidiarrheal drugs within one month of study entry.

Present intravenous drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - USC School of Medicine, Los Angeles, California
  - UCSD Med Ctr, San Diego, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Kaiser Permanente Med Ctr, San Francisco, California
  - San Mateo County Gen Hosp, San Mateo, California
  - Med Service, Miami, Florida
  - Emory Univ School of Medicine, Atlanta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Maine Med Ctr Med Clinics, Portland, Maine
  - Douglas Plesko, Boston, Massachusetts
  - Boston City Hosp, Boston, Massachusetts
  - Henry Ford Hosp, Detroit, Michigan
  - Univ of Missouri at Kansas City School of Medicine, Kansas City, Missouri
  - Mount Sinai Med Ctr, New York, New York
  - SUNY Stony Brook / Health Sciences Ctr, Stony Brook, New York
  - Einstein Med School, The Bronx, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Miriam Hosp / Family Healthcare Ctr at SSTAR, Providence, Rhode Island
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Infectious Disease Physicians Inc, Annandale, Virginia
  - Univ of Wisconsin School of Medicine, Madison, Wisconsin

REFERENCES:
- [Background] Romeu J, Miro JM, Mallolas J, Sirera G, Tortosa F, Clotet B. Sandostatin (SMS-201-995) in the long-term management of chronic diarrhea in AIDS patients. Int Conf AIDS. 1991 Jun 16-21;7(2):272 (abstract no WB2362)